CLINICAL TRIAL: NCT00698776
Title: Phase I/II Trial of Combination of Lenalidomide (Revlimid, LEN) and Autologous Mature Dendritic Cells Pulsed With α-galactosyl Ceramide (α-GalCer; KRN7000) in Myeloma
Brief Title: Combination of Lenalidomide and Autologous Mature Dendritic Cells Pulsed With KRN7000 in Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Kyowa Kirin Co., Ltd. (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0712003357
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Lenalidomide; KRN 7000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental): 10 mg/day in cohort 1, and 25 mg/day in cohort 2. LEN is administered orally in standard 21 day cycles starting one week before each DC injection and ending 14 days after each DC injection. All patients will receive a total of three cycles of LEN.
  Interventions: Drug: Lenalidomide; Biological: Monocyte derived DCs loaded with KRN7000

INTERVENTIONS:
Drug: Lenalidomide — 10 mg/day in cohort 1, and 25 mg/day in cohort 2. LEN is administered orally in standard 21 day cycles starting one week before each DC injection and ending 14 days after each DC injection. All patients will receive a total of three cycles of LEN.
  Other Names: Revlimid; LEN
Biological: Monocyte derived DCs loaded with KRN7000 — 10 million DCs injected intravenously
  Other Names: α-galactosyl-ceramide; α-GalCer

SUMMARY:
This is a single arm open label trial to test the tolerability of the combination of monocyte derived DCs loaded with KRN7000 (DC-KRN7000) and Lenalidomide (LEN) in patients with asymptomatic myeloma. Phase I component of the study will evaluate the optimal dose of LEN, with particular emphasis on safety. After an interim analysis of these data, a single dose level will be chosen for phase II component in additional patients.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated asymptomatic multiple myeloma
* Prior therapy: Patients cannot have received prior thalidomide, lenalidomide or corticosteroids for the intent of treating their myeloma. Prior corticosteroid use for the treatment of non-malignant disorders is permitted; concurrent use should be restricted to the equivalent of prednisone 10 mg per day or less. Prior radiation therapy for the treatment of solitary plasmacytoma is permitted, but more than 3 months should have elapsed from the last day of radiation.
* Measurable disease as defined by one of the following:

  * Serum monoclonal protein ≥1.0 g by protein electrophoresis
  * >200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Measurable soft tissue plasmacytoma.
  * ≥10% plasma cells as measured on the bone marrow aspirate or bone marrow biopsy.

    * Age ≥18 years.
    * ECOG Performance status 0, 1, or 2.
    * Willing to provide written informed consent.
    * All study participants must be registered into the mandatory RevAssistSM program, and be willing and able to comply with the requirements of RevAssistSM.
    * Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
    * Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

      (b) Laboratory inclusion criteria obtained ≤ 1 month prior to registration:
    * ANC ≥1500/μL
    * PLT ≥100,000/μL
    * Hemoglobin ≥8.0 g/dl
    * Creatinine ≤2.0 mg/dL (Any elevation above normal range should not be felt to be related to myeloma)

Exclusion Criteria:

* Solitary plasmacytoma.
* Uncontrolled infection.
* Another active malignancy.
* Immediate need for chemotherapy in the opinion of the treating physician.
* New York Heart Association classification III or IV.
* Existing ≥Grade 2 neuropathy.
* Any of the following:

  * Pregnant women
  * Nursing women
  * This study involves an agent that has known genotoxic, mutagenic and teratogenic effects. Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.)
  * Active systemic autoimmunity (e.g. systemic lupus erythematosus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of Dose Limiting Toxicities (DLTs) | upon completion of treatment

SECONDARY OUTCOMES:
Number of Natural Killer Cells(NKT)that make IFNγ in Vitro | upon completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Dhodapkar, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Richter J, Neparidze N, Zhang L, Nair S, Monesmith T, Sundaram R, Miesowicz F, Dhodapkar KM, Dhodapkar MV. Clinical regressions and broad immune activation following combination therapy targeting human NKT cells in myeloma. Blood. 2013 Jan 17;121(3):423-30. doi: 10.1182/blood-2012-06-435503. Epub 2012 Oct 24. PMID 23100308